CLINICAL TRIAL: NCT00790738
Title: Randomized Double-Blind Trial of Liothyronine (T3) Augmentation to Treatment as Usual vs Placebo For The Treatment of Bipolar Depression
Brief Title: Liothyronine (T3) for Bipolar Depression
Acronym: T3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Northwell Health (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Principal Investigator, Raphael Braga, MD, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 08-001
Record Dates: First submitted 2008-11-10; First posted 2008-11-13 (Estimated); Results first posted 2015-07-02 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: Depression; Bipolar Disorder
Keywords: bipolar disorder; depression; treatment; randomized controlled trial
MeSH Terms: conditions — Depression; Bipolar Disorder | interventions — Triiodothyronine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): liothyronine (T3)
  Interventions: Drug: Liothyronine (T3)
- 2 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Liothyronine (T3) — liothyronine (T3) up to 50 micrograms a day
  Other Names: cytomel (liothyronine)
  Arms: 1
Drug: placebo — placebo
  Arms: 2

SUMMARY:
This study evaluates the efficacy of the thyroid hormone T3 for depression in patients with bipolar disorder. In this study patients will be randomized to receive T3 or placebo.

DETAILED DESCRIPTION:
Bipolar affective disorder is a debilitating illness, and is characterized by depression episodes that dominates the longitudinal course and are most difficult to treat. Controlled trials with monotherapy mood stabilizers such as lithium and valproate show little to no efficacy and antidepressants may offer no additional efficacy. Recently there has been a growing interest in the use of quetiapine in bipolar depression. However, a successful treatment may take up to 8 weeks, and full remission is achieved in only 50% of patients. Thyroid hormone augmentation strategies have been used in unipolar depression with good results, but there is a paucity of its efficacy in bipolar depression (BD). To our knowledge there are no controlled studies regarding the efficacy of thyroid augmentation in BD. The present study proposes to evaluate the efficacy of T3 as an augmentation to treatment as usual in the treatment of BD. We plan to enroll patients with bipolar disorder I or II who are currently presenting with depressive symptoms. Patients will be randomized to 2 groups - liothyronine or placebo Results will provide information on the possible role of thyroid hormone augmentation in the treatment of patients with bipolar depression, and may contribute to alleviate the burden of this disabling condition.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-65;
2. DSM-IV diagnosis of BP I or BP II as per SCID;
3. Currently presenting with at least moderate levels of depression (HAM-D > 15;
4. Patient has to be on stable dose of at least one mood stabilizer (lithium, valproate, carbamazepine, lamotrigine, second generation antipsychotics) for at least 4 weeks as per history;
5. Antidepressants and/or additional mood stabilizers are allowed, but dose should be stable for at least 2 weeks;

Exclusion Criteria:

1. Evidence of acute mania or hypomania (as measured by CARS-M > 7);
2. Abnormal (outside of lab normal range) thyroid function tests;
3. Current thyroid hormone treatment;
4. Any medical condition considered a contraindication for treatment with T3 (i.e. history of myocardial infarction, cardiac arrhythmia, severe cardiac insufficiency, Autoimmune Thyroid Disease /Hashimoto's Thyroiditis as determined by anti-thyroid antibody testing, previous or current thyroid adenoma, hyperthyroidism);
5. EKG showing rhythm other than sinus or repolarization phase abnormalities;
6. Current alcohol or substance abuse or dependence in past month as per SCID;
7. Score of 3 or more on the suicide item of the HAM-D;
8. Females who are pregnant, breastfeeding, or of childbearing age and not using adequate birth control.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2008-07; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raphael J Braga, MD, Principal Investigator — The Zucker Hillside Hospital, North Shore - LIJHS
Locations (1):
- The Zucker Hillside Hospital, Glen Oaks, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Liothyronine (T3): liothyronine (T3)
  Liothyronine (T3): liothyronine (thyroid hormone T3) up to 50 micrograms a day.
Period: Overall Study
Arm/Group | Liothyronine (T3) | Placebo
Started | 5 | 6
Completed | 3 | 3
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Liothyronine (T3): liothyronine (T3)
  Liothyronine (T3): liothyronine (T3) up to 50 micrograms a day
- Total: Total of all reporting groups
Arm/Group | Liothyronine (T3) | Placebo | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (9.5) | 46.4 (5.9) | 45.2 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 1 | 5 | 6
Region of Enrollment [Number; unit: participants]
  United States | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Rating Scale for Depression Scores
Description: The Hamilton Rating Scale for Depression (HRSD) is a checklist of items ranked from 0-4 or 0-2, that was designed to measure the severity of depressive symptoms. The scale ranges from 0 to 50, and the following thresholds are used: very severe >23, severe 19-22, moderate 14-18, mild 8-13 and normal ≤7.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liothyronine (T3) | Placebo
Number analyzed (Participants) | 5 | 6
units on a scale | 3.50 (3.54) | 7.25 (5.44)

2. Secondary Outcome: Clinician-Administered Rating Scale for Mania
Description: The Clinician-Administered Rating Scale for Mania (CARS-M) contains 15 items rated from 0-5 or 0-6 on a Likert scale. It was developed to assess severity of manic symtoms. The scale ranges from 0 to 50, and the following thresholds are used: severe ≥26, moderate 16-25, mild 8-15 and normal ≤7.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liothyronine (T3) | Placebo
Number analyzed (Participants) | 5 | 6
units on a scale | 0.5 (0.71) | 2 (1.82)

3. Secondary Outcome: Clinical Global Impression Scores
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. At the time of rating patients are rated as: 1, normal, not at all ill; 2, borderline mentally ill; 3, mildly ill; 4, moderately ill; 5, markedly ill; 6, severely ill; or 7, extremely ill.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Liothyronine (T3) | Placebo
Number analyzed (Participants) | 5 | 6
units on a scale | 4 (0) | 3 (0)

ADVERSE EVENTS:
Arm/Group | Liothyronine (T3) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/5 | 1/6
Other Adverse Events (participants affected / at risk) | 4/5 | 4/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liothyronine (T3) (N=5) | Placebo (N=6)
Palpitation (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Liothyronine (T3) (N=5) | Placebo (N=6)
excitment (Nervous system disorders) | 0 (0) | 2 (2)
Malaise (General disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3) | 1 (1)
Hypersomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Drowsiness (Psychiatric disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 0 (0) | 1 (1)
Tinnitus (Nervous system disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Increased Appetite (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Despite several changes made in order to enhance recruitment during the study period, the study was markedly underpowered. Therefore, no definitive conclusions could be drawn from the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No